CLINICAL TRIAL: NCT02465255
Title: Sublingual Analgesia for Acute Abdominal Pain in Children. Ketorolac Versus Tramadol Versus Paracetamol, a Randomized, Control Trial
Brief Title: Sublingual Analgesia for Acute Abdominal Pain in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Luca Ronfani, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 22/13
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Abdominal Pain
Keywords: Acute Abdominal Pain; Sublingual Analgesia; Children; Ketorolac; Tramadol; Paracetamol; Analgesia
MeSH Terms: conditions — Abdominal Pain; Abdomen, Acute; Agnosia | interventions — Ketorolac; Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketorolac (Experimental): Ketorolac 0.5 mg/kg administrated by sublingual route
  Interventions: Drug: Ketorolac
- Tramadol (Active Comparator): Tramadol 2.0 mg/kg administrated by sublingual route
  Interventions: Drug: Tramadol
- Acetaminophen (paracetamol) (Active Comparator): Acetaminophen (paracetamol) 20.0 mg/kg administrated by sublingual route
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ketorolac
  Arms: Ketorolac
Drug: Tramadol
  Arms: Tramadol
Drug: Acetaminophen
  Arms: Acetaminophen (paracetamol)

SUMMARY:
Acute abdominal pain is a frequent symptom in children admitted to the emergency department . In the past the fear of masking a surgical condition has justified withholding analgesia in patients with acute abdominal pain. By the 2000s, some clinical trials established that opioid analgesia before surgical consultation does not affect diagnostic accuracy or outcome in children with acute abdominal pain. Despite this, acute abdominal pain is still undertreated in this setting. Published paediatric trials studied the effect of opioid analgesia administered by parenteral route or by mouth. To the best of our knowledge no study investigated the effectiveness of sublingual analgesia.

The purpose of this randomized controlled trial is to assess the effectiveness of three different drugs (ketorolac, tramadol, paracetamol), administered by the sublingual route, in children complaining of acute abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 18 years
* Emergency department admission for moderate to severe acute abdominal pain (VAS/NRS score >=6)
* Informed consent signed by parents or legal guardians

Exclusion Criteria:

* Known allergy or sensitivity to nonsteroidal anti-inflammatory drug, opioids or acetaminophen
* Use of analgesic drugs in the 8 hours before
* Clinical suspicion of abdominal pain due to fecal stasis
* Moderate or severe dehydration (weight loss of more than 5%)
* Known nephropathy, liver disease, metabolic or neurologic disease
* Thrombocytopenia or history of bleeding disease

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain Score | 120 minutes after drug administration
  Pain score evaluated with visual analogical scale (VAS) or Numeric Rating Scale (NRS) depending on child age

SECONDARY OUTCOMES:
Pain Score | 30 minutes after drug administration
  Pain score evaluated with visual analogical scale (VAS) or Numeric Rating Scale (NRS) depending on child age
Pain Score | 60 minutes after drug administration
  Pain score evaluated with visual analogical scale (VAS) or Numeric Rating Scale (NRS) depending on child age
Missed or delayed diagnosis of acute appendicitis or other abdominal pathology (i.e., pancreatitis) | 24 hours after drug administration
Missed or delayed diagnosis of acute appendicitis or other abdominal pathology (i.e., pancreatitis) | 48 hours after drug administration
Adverse events | up to 180 hours after the drug administration
  Presence of nausea, vomiting, diarrhea, headache, hyper- or hypotension, decreased excretion of urine, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Elena Neri, MD, Study Director — IRCCS Burlo Garofolo, Trieste, Italy; Giorgio Cozzi, MD, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy